CLINICAL TRIAL: NCT00857727
Title: Use of Dexmedetomidine for Emergence Delirium in Children Undergoing General Anesthesia for Endovascular Interventional Neuroradiologic Procedures
Brief Title: Use of Dexmedetomidine to Reduce Emergence Delirium Incident in Children
Acronym: DexPeds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dex Peds 08-088
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Results first posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Agitation; Anesthesia; Pediatrics
Keywords: Dexmedetomidine; Emergence Delirium; Agitation; Pediatric; Anesthesia
MeSH Terms: conditions — Psychomotor Agitation; Emergence Delirium | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug (Experimental): Dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- Control (Placebo Comparator): Normal Saline IV solution
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be dissolved in saline. An initial loading dose of 1.0 mg/kg given over 10 minutes followed by a continuous infusion at 0.4-0.7 mg/kg/hour. Beginning approximately one hour prior to end of surgery and continuing for one hour of recovery in the PACU and the PICU. This, the maximum dose for any one patient will be 2.4 mg/kg
  Other Names: Precedex
  Arms: Drug
Drug: Saline — Given by a continuous infusion
  Other Names: Phosphate buffered saline; PBS
  Arms: Control

SUMMARY:
Emergence delirium (ED) from general anesthesia posts risk and harm to pediatric population undergo general anesthesia. The purpose of the study is to compare the use of dexmedetomidine versus placebo in reducing the incidence and severity of ED in a pediatric neurosurgical population.

DETAILED DESCRIPTION:
Emergence delirium from general anesthesia is a common problem in the pediatric population with a reported incidence of up to 80%. In addition to being jarring to children and their parents, ED can cause significant physical harm, particularly to the surgical site. ED is also associated with accidental removal of surgical dressings and drains, intravenous and intra-arterial catheters, increased nursing care, extended recovery room stays, and delayed reunion with parents. Emergence delirium is especially associated with sevoflurane, the most commonly used inhalation anesthetic in pediatrics. At present, there is no single definition of pediatric ED because of its heterogeneous clinical presentation. It has been described as an acute phenomenon in which the child is irritable, uncompromising, uncooperative, incoherent, and inconsolably crying, moaning, kicking or thrashing. Typically, these children do not recognize or identify familiar objects or people, and often exhibit combative behavior. Although ED is a self-limiting phenomenon, it is especially dangerous in the interventional neuroradiologic patient whose femoral artery has been catheterized and must be kept immobile in the immediate post-operative period. These patients also have multiple intravenous and intra-arterial catheters which can be dislodged during an episode of ED. Numerous pharmacologic agents including benzodiazepines, opioids, ketamine, and clonidine, have been studied as prophylactic agents for ED but have met with varying success. Promising results with the α-2 adrenergic agonist clonidine, have spurred interest in a new α-2 adrenergic agonist, dexmedetomidine.

Dexmedetomidine is highly selective for the 2A subtype of the central presynaptic α-2 adrenergic receptor which is associated with sedation and analgesia. It is currently approved for use in adults as a sedative agent in intensive care units but has been used in myriad other ways for sedation. As a sedative, dexmedetomidine is unusual in that it does not depress respiratory drive because its actions are not mediated by the GABA-mimetic system. The quality of sedation produced by dexmedetomidine is unique, and has been described as "cooperative sedation," in which patients can interact with healthcare providers and follow verbal commands. This particular sedation profile permits a patient to be comfortably sedated, yet cooperate for an accurate neurological exam. The most extreme example of this is the awake craniotomy, in which a patient undergoes a neurological examination during surgery. In addition to being sedative, dexmedetomidine is also analgesic and suppresses shivering, making it especially useful in the perioperative period.

There have been studies suggesting a use for dexmedetomidine in ED yet none have examined its use in the pediatric neurosurgical population. Treatment of ED in pediatric neurosurgical patients involves balancing the need for smooth emergence with the need for accurate neurological exams. Benzodiazepines and opioids are currently used to treat ED but are long-acting, interfere with neurological exams, and carry the risks of respiratory depression, nausea, vomiting, and acute tolerance. Dexmedetomidine provides an alternative to current treatment modalities for ED, which does not interfere with neurological exams.

ELIGIBILITY:
Inclusion Criteria:

* Children age 6 months through 17 years of age undergoing interventional neuroradiologic procedures at our hospital under general anesthesia
* Patients classify as an ASA (American Society of Anesthesiologists) I-III
* Have not received anesthetic for over 30 days from previous procedures

Exclusion Criteria:

* Receiving digoxin therapy from the study
* Severe congestive heart failure or pulmonary hypertension requiring vasodilators
* Disease processes other than that associated with their intracranial pathology, such as hepatic or renal dysfunction

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2009-08; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jolie Narang, M.D., Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St Luke's-Roosevelt Hospital Center, New York, New York, United States

REFERENCES:
- [Background] Blaine Easley R, Brady KM, Tobias JD. Dexmedetomidine for the treatment of postanesthesia shivering in children. Paediatr Anaesth. 2007 Apr;17(4):341-6. doi: 10.1111/j.1460-9592.2006.02100.x. PMID 17359402
- [Background] Isik B, Arslan M, Tunga AD, Kurtipek O. Dexmedetomidine decreases emergence agitation in pediatric patients after sevoflurane anesthesia without surgery. Paediatr Anaesth. 2006 Jul;16(7):748-53. doi: 10.1111/j.1460-9592.2006.01845.x. PMID 16879517
- [Background] Guler G, Akin A, Tosun Z, Ors S, Esmaoglu A, Boyaci A. Single-dose dexmedetomidine reduces agitation and provides smooth extubation after pediatric adenotonsillectomy. Paediatr Anaesth. 2005 Sep;15(9):762-6. doi: 10.1111/j.1460-9592.2004.01541.x. PMID 16101707
- [Background] Ibacache ME, Munoz HR, Brandes V, Morales AL. Single-dose dexmedetomidine reduces agitation after sevoflurane anesthesia in children. Anesth Analg. 2004 Jan;98(1):60-63. doi: 10.1213/01.ANE.0000094947.20838.8E. PMID 14693585
- [Background] Walker J, Maccallum M, Fischer C, Kopcha R, Saylors R, McCall J. Sedation using dexmedetomidine in pediatric burn patients. J Burn Care Res. 2006 Mar-Apr;27(2):206-10. doi: 10.1097/01.BCR.0000200910.76019.CF. PMID 16566567

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 33 children undergoing general anesthesia for endovascular interventional procedures. 28 patients provided complete data sets.
Groups:
- Drug: Dexmedetomidine - An initial dose, given one hour prior to extubation of 1.0 µg/kg over 20 minutes, followed by a continuous infusion at 0.5 µg/kg/hour, continuing for 30 minutes following extubation.
- Control: Normal Saline IV solution - Given by a continuous infusion
Period: Overall Study
Arm/Group | Drug | Control
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug | Control | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.2 (2.6) | 4.2 (2.7) | 4.7 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Emergence Delirium
Description: Emergence Delirium (ED) during the 15-45min. post-op period as assessed by the Cole Score. (Cole Score 3-5 = ED). The Cole Scale is an ordinal ranking of ED (1=sleeping; 2=awake, calm; 3=irritable, crying; 4=inconsolable, crying; 5=severe restlessness, disorientation).
Time Frame: 15-45 minutes post-op
Measure: Number; unit: participants
Arm/Group | Drug | Control
Number analyzed (Participants) | 14 | 14
participants
  ED | 1 | 7
  No ED | 13 | 7

2. Secondary Outcome: Vital Signs (Heart Rate, Blood Pressure, Respiratory Rate and Pulse Oximetry) Will be Continuously Monitored in the PICU
Description: Vital signs were not collected as part of research study.
Time Frame: 24 hours
Population: data were not collected
Arm/Group | Drug | Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Weight
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Drug | Control
Number analyzed (Participants) | 14 | 14
kg | 21.8 (7.3) | 18.5 (8.1)

4. Secondary Outcome: Length of Anesthesia
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Drug | Control
Number analyzed (Participants) | 14 | 14
minutes | 199 (71) | 215 (156)

5. Secondary Outcome: Length of Surgery
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Drug | Control
Number analyzed (Participants) | 14 | 14
minutes | 58 (43) | 86 (149)

6. Secondary Outcome: Total Study Drug
Description: Total Study Drug used
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mcg/kg
Arm/Group | Drug | Control
Number analyzed (Participants) | 14 | 14
mcg/kg | 1.55 (0.32) | 1.43 (0.32)

7. Secondary Outcome: Total Sevoflurane
Description: Total Drug used
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Drug | Control
Number analyzed (Participants) | 14 | 14
ml/kg | 3.67 (1.38) | 6.80 (7.81)

8. Secondary Outcome: Total Propofol
Description: Total Drug used
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Drug | Control
Number analyzed (Participants) | 14 | 14
mg/kg | 2.11 (1.28) | 2.41 (1.36)

9. Secondary Outcome: Total Fentanyl
Description: Total Drug used
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mcg/kg
Arm/Group | Drug | Control
Number analyzed (Participants) | 14 | 14
mcg/kg | 2.33 (0.79) | 2.36 (0.99)

ADVERSE EVENTS:
Description: Two adverse events were noted requiring unblinding
Arm/Group | Drug | Control
Serious Adverse Events (participants affected / at risk) | 1/14 | 1/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug (N=14) | Control (N=14)
Severe bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Excessive sedation (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Methodology used cannot determine whether undescribed prolonged effect of DEX is related to the DEX or to increased activity levels in the placebo group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes